CLINICAL TRIAL: NCT06326008
Title: Safety, Tolerability and Pharmacokinetics of Donor-derived CD19 CAR Therapy Bridged Allogeneic Haematopoietic Stem Cell Transplantation and Sequential Donor-derived CD22 CAR Therapy in Refractory or Relapsed B Cell Acute Lymphoblastic Leukemia: a Clinical Trial
Brief Title: Safety, Tolerability, and Pharmacokinetics of Donor-derived CD19 CAR Therapy Bridged Allo-HSCT and Sequential Donor-derived CD22 CAR Therapy for r/r B-ALL: a Clinical Trial
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Responsible Party: Principal Investigator, Jing Pan, Director of Dept of Hemato-Oncology and Immunotherapy, Beijing GoBroad Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJGBYY-IIT-LCYJ-2023-002
Record Dates: First submitted 2024-03-10; First posted 2024-03-22 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; Acute Lymphoblastic Leukemia, in Relapse
MeSH Terms: conditions — Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm-1 (Experimental): Participants receive donor-derived CD19 CAR therapy bridged Allo-HSCT and sequential donor-derived CD22 CAR therapy
  Interventions: Drug: Donor-derived CD19 CAR Therapy Bridged Allo-HSCT and Sequential Donor-derived CD22 CAR Therapy

INTERVENTIONS:
Drug: Donor-derived CD19 CAR Therapy Bridged Allo-HSCT and Sequential Donor-derived CD22 CAR Therapy — Peripheral blood mononuclear cells for the production of CD19 CAR T cells and CD22 CAR T cells are collected from donors and haematopoietic stem cells are collected from donors.

SUMMARY:
This is an investigator-initiated, single-arm, open-label, non-randomised phase I clinical study. The objective of this trial is to evaluate the safety, tolerability and pharmacokinetics of donor-derived CD19 CAR Therapy bridged Allo-HSCT and sequential donor-derived CD22 CAR Therapy for r/r B-ALL and to explore the efficacy of this therapy preliminarily. The primary endpoints are incidence and type of dose-limiting toxicity (DLT) within 28 days (i.e., 43 days after donor-derived CD19 CAR T-cell infusion) after donor-derived CD19 CAR T-cell therapy bridged allogeneic haematopoietic stem cell transplantation; total number, incidence and severity of adverse events from donor-derived CD19 CAR T cell infusion back to 30 days after donor-derived CD22 CAR T cell infusion (i.e., within 120 days of donor-derived CD19 CAR T cell infusion). The secondary endpoints are total number, incidence and severity of adverse events from 120 days to 2 years after donor-derived CD19 CAR T-cell infusion; ORR(CR+CRi) on days 45, 90, 120; duration of response(DOR), event-free survival(EFS), overall survival(OS); pharmacokinetics characteristics. The trial plan to enroll 3~12 cases in dose escalation phase and 36 cases in dose expansion phase.

ELIGIBILITY:
Inclusion Criteria:

- Patients will be enrolled only if they meet all the inclusion criteria.

1. Patients with relapsed or refractory CD19+/CD22+ (FCM >95%) B-cell acute lymphoblastic leukaemia who have progressed despite or are intolerant to all standard therapies, including, but not limited to, immunotherapies such as Blinatumomab (BITE), Tyrosine kinase inhibitors (TKI), CAR T-cell therapy, etc.; Currently available therapies have a limited prognosis and there are no available curative treatment options (e.g., HSCT or chemotherapy);
2. Peripheral blood tumour burden ≥60% or severe peripheral blood cytopenia, unsuitable/unable to collect autologous lymphocytes;
3. 1 to 18 years old;
4. Patient's expected survival time ≥ 60 days;
5. Physical status: ECOG score 0-2;
6. Availability of allogeneic donors (HLA-identical or HLA-haploidentical) DSA-negative for collection of peripheral blood mononuclear cells and peripheral blood stem cells;
7. Sign an informed consent form during the screening period. Pediatric patients under 8~18 years of age need to have sufficient awareness to voluntarily sign an informed consent form, and their legal representatives (guardians) also need to voluntarily sign an informed consent form; pediatric patients aged 1~7 years can only be recruited after their legal guardians have voluntarily signed an informed consent form.

Exclusion Criteria:

* Patients who meet any of the following criteria are not eligible for enrolment.

  1. Patients who have received previous haematopoietic stem cell transplantation (including peripheral blood haematopoietic stem cell transplantation and bone marrow haematopoietic stem cell transplantation);
  2. Intracranial hypertension or cerebral impaired consciousness;
  3. Symptomatic heart failure or severe cardiac arrhythmia;
  4. Symptoms of severe respiratory failure;
  5. With other types of malignant tumours;
  6. Diffuse intravascular coagulation;
  7. Serum creatinine and/or urea nitrogen ≥ 1.5 times the normal value;
  8. Suffering from sepsis or other uncontrollable infections;
  9. Suffering from uncontrollable diabetes mellitus;
  10. Severe mental disorders;
  11. Have significant intracranial lesions on cranial MRI (excluding intracranial masses caused by central nervous system leukaemia);
  12. Have organ transplant history;
  13. Female patients (patients of childbearing potential) with positive blood HCG test;
  14. Hepatitis (including Hepatitis B and Hepatitis C) and positive screening for AIDS and syphilis;
  15. No allogeneic donor suitable for collection of peripheral blood lymphocytes and haematopoietic stem cells.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Within 43 days of donor-derived CD19 CAR T-cell infusion
  Incidence and type of dose-limiting toxicity (DLT) within 28 days (i.e., 43 days after donor-derived CD19 CAR T-cell infusion) after donor-derived CD19 CAR T-cell therapy bridging allogeneic haematopoietic stem cell transplantation will be recorded.
Adverse events (AEs) | Within 120 days of donor-derived CD19 CAR T-cell infusion
  Total number, incidence and severity of adverse events (AEs) from the time of donor-derived CD19 CAR T cell infusion back to 30 days after donor-derived CD22 CAR T cell infusion (i.e., within 120 days of donor-derived CD19 CAR T-cell infusion) will be recorded.

SECONDARY OUTCOMES:
Long-term Adverse events (AEs) | From 120 days to 2 years after donor-derived CD19 CAR T-cell infusion
  Total number, incidence and severity of AEs from 120 days to 2 years after donor-derived CD19 CAR T-cell infusion will be recorded.
Objective response rate(ORR) | day 30, day 45, day 90
  Objective response rate (ORR) at day 30, day 45, day 90 as determined by the National Comprehensive Cancer Network (NCCN) GuidelinesVersion 3.2023 of Acute Lymphoblastic Leukemia.
Duration of response (DOR) | Up to 2 years
  DOR is defined as the date when CR or CRi response criteria are first met to the date of relapse or death caused by ALL in the absence of documented relapse.
Event-free survival (EFS) | Up to 2 years
  EFS is defined as the time from donor-derived CD19 CAR T-cell infusion to the occurrence of any event, which includes disease progression, discontinuation of therapy for any reason, or death.
Overall survival (OS) | Up to 2 years
  OS is defined as the time from the infusion of donor-derived CD19 CAR T cells until death due to any cause.
The persistence of CD19/CD22 CAR T cells. | Up to 2 years
  The persistence of CD19/CD22 CAR T cells in cerebral spinal fluid (CSF) and peripheral blood will be detected by flowcytometry and qPCR after CD19/CD22 CAR T cells infusion.
The Maximum concentration (Cmax) of CD19/CD22 CAR T cells. | Up to 2 years
  The Maximum concentration (Cmax) of CD19/CD22 CAR T cells will be recorded.
The time to maximum plasma concentration (Tmax) of CD19/CD22 CAR T cells. | Up to 2 years
  The time to maximum plasma concentration (Tmax) of CD19/CD22 CAR T cells will be recorded.